CLINICAL TRIAL: NCT04547868
Title: Can Coffee/Caffeine Improve Post-Operative Gastrointestinal Recovery? A Vanguard Randomized Controlled Trial
Brief Title: Can Coffee/Caffeine Improve Post-Operative Gastrointestinal Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Paul Karanicolas, Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO Project ID: 2121
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Ileus; Caffeine
Keywords: Postoperative gastrointestinal recovery; Gastrointestinal motility; Coffee
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Intervention Model Description: Pragmatic, multicentre, open-label, three-arm parallel group Vanguard feasibility randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coffee (Experimental): Caffeinated coffee beverage
  Interventions: Other: Coffee
- Decaffeinated coffee (Active Comparator): Decaffeinated coffee beverage
  Interventions: Other: Decaffeinated Coffee
- Warm water (Placebo Comparator): Warm water beverage
  Interventions: Other: Warm water

INTERVENTIONS:
Other: Coffee — Once the surgical team deems it appropriate to begin a clear liquid diet (in the post-operative period), approximately one cup of coffee will be provided to the patient three times daily. Additives such as cream, milk, sweetener and sugar, will be permitted. The intervention(s) will continue until a change is required as per the treating team or until hospital discharge. Patients will be asked to avoid any additional caffeine intake, such as tea, for the duration of the trial. If a patient receives an NG tube or is placed NPO by the treating team, the intervention will be halted and restarted once a clear liquid diet is restarted. All other aspects of the patients' care will be at the discretion of the treating team as per their standard practices.
  Arms: Coffee
Other: Decaffeinated Coffee — Once the surgical team deems it appropriate to begin a clear liquid diet (in the post-operative period), approximately one cup of decaffeinated coffee will be provided to the patient three times daily. Additives such as cream, milk, sweetener and sugar, will be permitted. The intervention(s) will continue until a change is required as per the treating team or until hospital discharge. Patients will be asked to avoid any additional caffeine intake, such as tea, for the duration of the trial. If a patient receives an NG tube or is placed NPO by the treating team, the intervention will be halted and restarted once a clear liquid diet is restarted. All other aspects of the patients' care will be at the discretion of the treating team as per their standard practices.
  Arms: Decaffeinated coffee
Other: Warm water — Once the surgical team deems it appropriate to begin a clear liquid diet (in the post-operative period), approximately one cup of warm water will be provided to the patient three times daily. Additives such as cream, milk, sweetener and sugar, will be permitted. The intervention(s) will continue until a change is required as per the treating team or until hospital discharge. Patients will be asked to avoid any additional caffeine intake, such as tea, for the duration of the trial. If a patient receives an NG tube or is placed NPO by the treating team, the intervention will be halted and restarted once a clear liquid diet is restarted. All other aspects of the patients' care will be at the discretion of the treating team as per their standard practices.
  Arms: Warm water

SUMMARY:
Disruption of the normal gastrointestinal (GI) motility is a well-known consequence of major surgery. The pathophysiology behind this phenomenon is not fully understood but involves the autonomic nervous system as well as a systemic stress response to surgery. A number of factors interfere with GI motor activity, such as the direct manipulation of intestines during surgery and the use of opioid analgesia. Post-operative ileus (POI) refers to a delay in regaining GI motility beyond the anticipated normal duration of time. Signs and symptoms include nausea, vomiting, abdominal distention, the absence of flatus or stool in the preceding 24 hours, and/or an inability to tolerate oral intake. The incidence of POI in abdominal surgery is estimated to be approximately 10%-30%. Beyond increased patient discomfort and distress, the development of POI is associated with increased healthcare costs.

Coffee is a popular beverage: two thirds of Canadians are coffee drinkers, averaging approximately 3.2 cups per day. Coffee is composed of hundreds of chemicals, many with demonstrated pharmacologic effects. The most well-known of these compounds is caffeine, known to exert a stimulatory effect on the cardiovascular and nervous system. A recent systematic review of 7 randomized controlled trials (N=606 colorectal and gynecology surgical patients) determined that the consumption of coffee reduced the time of several measures of GI recovery, such as time to tolerance of food, without any increased rate of complications or adverse events although overall, the evidence was graded as low to moderate certainty, and further confirmatory studies are needed. In this trial, patients aged 18 years or higher who undergo laparoscopic or open abdominal surgery, with an estimated length of stay > 24 hours will be randomized to receive approximately one cup of either coffee, decaffeinated coffee, or warm water, three times daily. This trial will be conducted under the IMPACTS (Innovative, Multicentre, Patient-centred Approach to Clinical Trials in Surgery) program umbrella and will follow IMPACTS methodology. For the Vanguard trial, the aim is to determine the feasibility of conducting a definitive trial. Future outcomes of interest include: time to first flatus, time to first bowel movement, placement of an NG tube, length of stay in hospital, 30-day mortality, and 30-day postoperative complications.

DETAILED DESCRIPTION:
Background/rationale: The development of POI is a common complication of surgery that is detrimental to patient well-being and ultimately leads to significant healthcare costs. Coffee is a popular drink among Canadians and appears to exert a positive effect on GI motility. This beverage may provide an inexpensive, easily administered and well-tolerated intervention to accelerate post-operative GI recovery, and thus reduce POI. The current literature, while promising, is insufficient and merits further investigation in the form of a high-quality randomized controlled trial.

Objectives: Before embarking on a definitive RCT, this pilot trial has five specific feasibility objectives:

1. To assess our ability to accrue patients using the IMPACTS Program platform, at multiple institutions, over the course of one year.
2. To assess our ability to adaptively randomize patients and deliver the randomized assignment using the IMPACTS Program platform, over the course of one year.
3. To assess our ability to collect complete data directly from participants (patients and clinicians) on time to first flatus and time to first bowel movement over the course of one year.
4. To examine our ability to carry out data linkages using the IMPACTS Program platform over the course of one year.
5. To estimate the change in time to first flatus to inform the sample size calculation for the definitive trial.

Study design: This is a multicentre, pragmatic, 3-arm parallel group Vanguard feasibility randomized controlled trial. Patients will be randomly assigned to consume coffee, decaffeinated coffee, or warm water. If feasibility is demonstrated during the pilot trial, we will plan to conduct a definitive trial. If there are only minimal changes to the protocol, we will include data from the pilot phase into the definitive trial analysis (i.e. a Vanguard design).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Planned elective laparoscopic or open abdominal surgery
* Patient is scheduled to remain in hospital for at least one night, post-operatively

Exclusion Criteria:

* Known intolerance to coffee or caffeine
* Unwilling to stop current caffeine consumption (coffee or tea) during trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-21 (Actual)

PRIMARY OUTCOMES:
Assessment of accrual | 1 year
  Average number of patients enrolled per month across the 3 sites for the trial: feasible if 10 or more
Ability to deliver intervention patient is randomized to receive | 1 year
  Feasible if > 90% of patients receive the correct intervention
Ability to collect complete data for patient-reported outcomes | 1 year
  Feasible if > 80% of data is collected
Ability to link data from patient-reported outcome measures with Institute for Clinical/Evaluative Sciences and National Surgical Quality Improvement Program datasets | 1 year
  Feasible if linkage is possible in > 90% of patients
Measurement of baseline data | 1 year
  1. Median number of hours until flatus in control group
  2. Median number of hours until flatus in coffee and decaffeinated coffee groups

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - North York General Hospital, North York, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No